CLINICAL TRIAL: NCT00091507
Title: Immediate Myocardial Metabolic Enhancement During Initial Assessment and Treatment in Emergency Care Trial
Brief Title: IMMEDIATE Trial - Out of Hospital Administration of Glucose, Insulin and Potassium.
Acronym: IMMEDIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 165; U01HL077826 (NIH); U01HL077823 (NIH); U01HL077822 (NIH); U01HL077821 (NIH)
Record Dates: First submitted 2004-09-09; First posted 2004-09-13 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Angina, Unstable; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Heart Failure, Congestive
Keywords: Acute Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Myocardial Infarction; Heart Failure; Acute Coronary Syndrome | interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 -- GIK (Experimental): GIK = glucose-insulin-potassium; In one-liter: Dextrose 30% + 80 mEq Potassium Chloride + 50 units Regular Insulin; infused at 1.5 ml/kg/hour for a total of 12 hours.
  Interventions: Drug: GIK
- 2 -- Placebo (Placebo Comparator): Dextrose 5%, infused at 1.5 ml/kg/hour for total of 12 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GIK — Intravenous solution, 1.5ml/kg/hour, continuous infusion for total of 12 hours.
  Other Names: Glucose-Insulin Potassium
  Arms: 1 -- GIK
Drug: Placebo — Intravenous solution of Dextrose 5 percent at 1.5 ml/kg/hour for a total of 12 hours.
  Other Names: Dextrose 5%
  Arms: 2 -- Placebo

SUMMARY:
The purpose of this study is to test the impact of pharmacological myocardial metabolic support, in the form of intravenous (IV) glucose, insulin and potassium (GIK), for the treatment of patients with threatened or established acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
BACKGROUND:

Basic and clinical research suggests intravenous GIK metabolic myocardial support reduces ischemia-induced arrhythmias, progression from unstable angina pectoris (UAP) to acute myocardial infarction (AMI), myocardial infarction (MI) size, and mortality. Also, for ST elevation MI (STEMI), GIK may prolong time of benefit of coronary reperfusion. These effects should reduce short- and long-term mortality from ACS, including AMI and UAP, and the propensity for heart failure (HF). These benefits are related to the earliness of ACS, when both risk and opportunity to save lives are highest.

DESIGN NARRATIVE:

This is a randomized, placebo-controlled, double-blinded, multicenter clinical trial of IMMEDIATE GIK as early as possible in ACS in the prehospital emergency medical service (EMS) setting. Distinct from prior and ongoing GIK trials, this will test GIK for all ACS rather than only for AMI or STEMI in prehospital EMS. The primary hypothesis is that early GIK will prevent or reduce the size of acute myocardial infarction. Major secondary hypotheses posit GIK will reduce mortality (30 days and 1 year), reduce pre- or in-hospital cardiac arrest and the propensity for heart failure. Other hypotheses address mechanisms of these effects.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of threatened or established AMI including but not limited to:

  1. Chest pain, discomfort, or tightness
  2. Arm or shoulder pain
  3. Jaw pain
  4. Epigastric discomfort
  5. Shortness of breath
* 12-lead electrocardiogram (ECG) with two or more contiguous leads with ST elevation greater than 1 mm, ST depression greater than 0.5 mm, T wave inversion or other T wave abnormalities (hyperacute T waves), or left bundle branch block (not known to be old). Identification aided by the acute cardiac ischemia time-insensitive predictive instrument (ACI-TIPI)and thrombolytic predictive instrument (TPI) decision support software (ACI-TIPI >= 75% and TPI detection of suspected STEMI).

Exclusion Criteria:

* End-stage kidney failure requiring dialysis
* Rales present more than halfway up the back
* Unable to comply with the requirements of the study
* Incarcerated
* Known to be pregnant

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 911 (Actual)
Dates: Start 2006-11; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Selker, MD, MSPH, Study Chair — Tufts Medical Center, Trial Coordinating Center; Ralph D'Agostino, PhD, Principal Investigator — Tufts Medical Center, Data Coordinating Center; James Udelson, MD, Principal Investigator — Tufts Medical Center, LV Core Lab
Locations (13):
- United States (13):
  - Anchorage Site, Anchorage, Alaska
  - New Haven Site, New Haven, Connecticut
  - Macon Site, Macon, Georgia
  - Brockton Site, Brockton, Massachusetts
  - Concord Site, Concord, Massachusetts
  - St. Paul Site, Saint Paul, Minnesota
  - Albuquerque Site, Albuquerque, New Mexico
  - Hershey Site, Hershey, Pennsylvania
  - Sioux Falls Site, Sioux Falls, South Dakota
  - Dallas Site, Dallas, Texas
  - El Paso Site, El Paso, Texas
  - Bellingham Site, Bellingham, Washington
  - Milwaukee Site, Milwaukee, Wisconsin

REFERENCES:
- [Background] Selker HP, Beshansky JR, Ruthazer R, Sheehan PR, Sayah AJ, Atkins JM, Aufderheide TP, Pirrallo RG, D'Agostino RB, Massaro JM, Griffith JL. Emergency medical service predictive instrument-aided diagnosis and treatment of acute coronary syndromes and ST-segment elevation myocardial infarction in the IMMEDIATE trial. Prehosp Emerg Care. 2011 Apr-Jun;15(2):139-48. doi: 10.3109/10903127.2010.545478. PMID 21366431
- [Background] Selker HP, Beshansky JR, Griffith JL, D'Agostino RB, Massaro JM, Udelson JE, Rashba EJ, Ruthazer R, Sheehan PR, Desvigne-Nickens P, Rosenberg YD, Atkins JM, Sayah AJ, Aufderheide TP, Rackley CE, Opie LH, Lambrew CT, Cobb LA, Macleod BA, Ingwall JS, Zalenski RJ, Apstein CS. Study design for the Immediate Myocardial Metabolic Enhancement During Initial Assessment and Treatment in Emergency Care (IMMEDIATE) Trial: A double-blind randomized controlled trial of intravenous glucose, insulin, and potassium for acute coronary syndromes in emergency medical services. Am Heart J. 2012 Mar;163(3):315-22. doi: 10.1016/j.ahj.2012.02.002. PMID 22424000
- [Background] Ellis KL, Zhou Y, Rodriguez-Murillo L, Beshansky JR, Ainehsazan E, Selker HP, Huggins GS, Cupples LA, Peter I. Common variants associated with changes in levels of circulating free fatty acids after administration of glucose-insulin-potassium (GIK) therapy in the IMMEDIATE trial. Pharmacogenomics J. 2017 Jan;17(1):76-83. doi: 10.1038/tpj.2015.84. Epub 2015 Dec 8. PMID 26644202
- [Background] Ellis KL, Zhou Y, Beshansky JR, Ainehsazan E, Selker HP, Cupples LA, Huggins GS, Peter I. Genetic modifiers of response to glucose-insulin-potassium (GIK) infusion in acute coronary syndromes and associations with clinical outcomes in the IMMEDIATE trial. Pharmacogenomics J. 2015 Dec;15(6):488-95. doi: 10.1038/tpj.2015.10. Epub 2015 Mar 17. PMID 25778467
- [Background] Alkofide H, Huggins GS, Beshansky JR, Ruthazer R, Peter I, Ray M, Mukherjee JT, Selker HP. C-Reactive protein reactions to glucose-insulin-potassium infusion and relations to infarct size in patients with acute coronary syndromes. BMC Cardiovasc Disord. 2015 Dec 3;15:163. doi: 10.1186/s12872-015-0153-7. PMID 26631004
- [Background] Alkofide H, Huggins GS, Ruthazer R, Beshansky JR, Selker HP. Serum adiponectin levels in patients with acute coronary syndromes: Serial changes and relation to infarct size. Diab Vasc Dis Res. 2015 Nov;12(6):411-9. doi: 10.1177/1479164115592638. Epub 2015 Jul 20. PMID 26193887
- [Result] Selker HP, Beshansky JR, Sheehan PR, Massaro JM, Griffith JL, D'Agostino RB, Ruthazer R, Atkins JM, Sayah AJ, Levy MK, Richards ME, Aufderheide TP, Braude DA, Pirrallo RG, Doyle DD, Frascone RJ, Kosiak DJ, Leaming JM, Van Gelder CM, Walter GP, Wayne MA, Woolard RH, Opie LH, Rackley CE, Apstein CS, Udelson JE. Out-of-hospital administration of intravenous glucose-insulin-potassium in patients with suspected acute coronary syndromes: the IMMEDIATE randomized controlled trial. JAMA. 2012 May 9;307(18):1925-33. doi: 10.1001/jama.2012.426. Epub 2012 Mar 27. PMID 22452807
- [Derived] Selker HP, Udelson JE, Massaro JM, Ruthazer R, D'Agostino RB, Griffith JL, Sheehan PR, Desvigne-Nickens P, Rosenberg Y, Tian X, Vickery EM, Atkins JM, Aufderheide TP, Sayah AJ, Pirrallo RG, Levy MK, Richards ME, Braude DA, Doyle DD, Frascone RJ, Kosiak DJ, Leaming JM, Van Gelder CM, Walter GP, Wayne MA, Woolard RH, Beshansky JR. One-year outcomes of out-of-hospital administration of intravenous glucose, insulin, and potassium (GIK) in patients with suspected acute coronary syndromes (from the IMMEDIATE [Immediate Myocardial Metabolic Enhancement During Initial Assessment and Treatment in Emergency Care] Trial). Am J Cardiol. 2014 May 15;113(10):1599-605. doi: 10.1016/j.amjcard.2014.02.010. Epub 2014 Mar 1. PMID 24792735
- [Derived] Beshansky JR, Sheehan PR, Klima KJ, Hadar N, Vickery EM, Selker HP. A community consultation survey to evaluate support for and success of the IMMEDIATE trial. Clin Trials. 2014 Apr;11(2):178-86. doi: 10.1177/1740774514526476. PMID 24686107
- [Derived] Sullivan AL, Beshansky JR, Ruthazer R, Murman DH, Mader TJ, Selker HP. Factors associated with longer time to treatment for patients with suspected acute coronary syndromes: a cohort study. Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):86-94. doi: 10.1161/CIRCOUTCOMES.113.000396. Epub 2014 Jan 14. PMID 24425697

RESULTS

PARTICIPANT FLOW:
Groups:
- GIK --: GIK = glucose-insulin-potassium
- Placebo: Dextrose 5%
Period: Overall Study
Arm/Group | GIK -- | Placebo
Started | 432 | 479
Completed | 411 | 460
Not Completed | 21 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GIK -- | Placebo | Total
Number analyzed (Participants) | 432 | 479 | 911
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (13.9) | 63.3 (14.1) | 63.6 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 146 | 265
  Male | 313 | 333 | 646
Region of Enrollment [Number; unit: participants]
  United States | 432 | 479 | 911

OUTCOME MEASURES:

1. Primary Outcome: Progression of Acute Coronary Syndrome to Myocardial Infarction
Description: Outcome for all participants during the first 24 hours of hospitalization; evidence of myocardial infarction is determined by ECG and biomarker results.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | GIK -- | Placebo
Number analyzed (Participants) | 411 | 460
participants | 200 | 242
Statistical Analysis 1: Comparison: GIK -- vs Placebo; Test type: Superiority or Other; p = 0.28, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.66 to 1.13]

2. Secondary Outcome: Cardiac Arrest
Description: Outcome for all participants who had a cardiac arrest from initial contact in the prehospital setting through their subsequent hospitalization.
Time Frame: 1 to 18 hours (From prehospital setting through hospitalization.)
Measure: Number; unit: participants
Arm/Group | GIK -- | Placebo
Number analyzed (Participants) | 411 | 460
participants | 15 | 29
Statistical Analysis 1: Comparison: GIK -- vs Placebo; Test type: Superiority or Other; p = 0.08, Regression, Logistic; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.30 to 1.07]

3. Secondary Outcome: Heart Failure or Death
Description: Outcome for all participants (composite of re-hospitalization for heart failure or death within 30 days)
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | GIK -- | Placebo
Number analyzed (Participants) | 411 | 460
participants | 23 | 35
Statistical Analysis 1: Comparison: GIK -- vs Placebo; Test type: Superiority or Other; p = 0.24, Regression, Logistic; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.43 to 1.23]

4. Secondary Outcome: Mortality
Description: Outcome for all participants (mortality at 30 days).
Time Frame: 30 days
Population: 30 day mortality.
Measure: Number; unit: participants
Arm/Group | GIK -- | Placebo
Number analyzed (Participants) | 411 | 460
participants | 18 | 28
Statistical Analysis 1: Comparison: GIK -- vs Placebo; Test type: Superiority or Other; p = 0.27, Regression, Logistic; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.40 to 1.29]

5. Secondary Outcome: Cardiac Arrest or Acute Mortality
Description: Outcome for all participants (composite of cardiac arrest or acute mortality)
Time Frame: Prehospital setting through hospitalization
Measure: Number; unit: participants
Arm/Group | GIK -- | Placebo
Number analyzed (Participants) | 411 | 460
participants | 18 | 40
Statistical Analysis 1: Comparison: GIK -- vs Placebo; Test type: Superiority or Other; p = 0.01, Regression, Logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.27 to 0.85]

ADVERSE EVENTS:
Arm/Group | GIK -- | Placebo
Serious Adverse Events (participants affected / at risk) | 28/411 | 41/460
Other Adverse Events (participants affected / at risk) | 295/411 | 199/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIK -- (N=411) | Placebo (N=460)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 4 (4) | 13 (13)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 4 (4) | 10 (10)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 6 (6) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 6 (6)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Hyperkaelemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIK -- (N=411) | Placebo (N=460)
Cardiac failure congestive (Cardiac disorders) | 19 (19) | 17 (17)
Ventricular extrasystoles (Cardiac disorders) | 25 (25) | 32 (32)
Ventricular tachycardia (Cardiac disorders) | 24 (24) | 30 (30)
Hyperglycaemia (Endocrine disorders) | 147 (147) | 66 (66)
Hypoglycaemia (Endocrine disorders) | 35 (35) | 3 (3)
Injection site reaction (General disorders) | 58 (58) | 10 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 27 (27) | 13 (13)
Hypotension (Vascular disorders) | 29 (29) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No